CLINICAL TRIAL: NCT06048926
Title: A Randomized, Double-blind, Parallel-controlled, Multicenter Phase III Clinical Study
Brief Title: Carrelizumab Combined With Concurrent Radiotherapy and Chemotherapy for Unresectable Esophageal Squamous Cell Carcinoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GXL-004
Record Dates: First submitted 2023-03-16; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Carrelizumab; Concurrent chemoradiotherapy; Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab; Paclitaxel; Drug Therapy; Cisplatin; Chemoradiotherapy; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: carrelizumab in combination with concurrent chemoradiotherapy (Experimental): Study drugs were administered intravenously on the first day of each cycle. Administered sequentially: carrelizumab, 200mg/time, paclitaxel, 50mg/m2, cisplatin, 25mg/m2, chemotherapy once a week, a total of 5 doses, carrelizumab every three weeks until PD or intolerable, up to 2 years, simultaneous radiotherapy at the first dose, the total dose of radiotherapy is 50.4Gy, completed in 28 divided doses, 1.8Gy each time, 5 times a week.
  Interventions: Drug: Carrelizumab; Drug: Paclitaxel injection; Drug: Cisplatin; Radiation: Concurrent chemoradiotherapy
- Control group: placebo-resistant in combination with chemoradiotherapy (Placebo Comparator): Placebo: 200 mg intravenously given with Q3W until PD or intolerable, carrelizumab/placebo for up to 2 years.
  Paclitaxel: 50mg/m2, iv, D1, 8, 15, 22, 29, once a week, a total of 5 times. cisplatin: 25mg/m2,iv, D1, 8, 15, 22, 29, once a week, a total of 5 doses. Radiotherapy: total dose of 50.4 Gy, completed in 28 divided doses of 1.8 Gy each time, 5 times a week.
  Interventions: Drug: Paclitaxel injection; Drug: Cisplatin; Radiation: Concurrent chemoradiotherapy

INTERVENTIONS:
Drug: Carrelizumab — 200 mg/time, iv, Q3W
  Other Names: Erica
  Arms: Experimental group: carrelizumab in combination with concurrent chemoradiotherapy
Drug: Paclitaxel injection — 50mg/m2,iv, D1, 8, 15, 22, 29, once a week, a total of 5 times
  Other Names: chemotherapy
Drug: Cisplatin — 25mg/m2，iv， D1、8、15、22、29，once a week, a total of 5 times
  Other Names: chemotherapy
Radiation: Concurrent chemoradiotherapy — Radiotherapy was given simultaneously at the time of the first dose, and the total dose of radiotherapy was 50.4 Gy, which was completed in 28 divided doses of 1.8 Gy each time, 5 times a week.
  Other Names: Radiotherapy

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multicenter phase III clinical study to evaluate the efficacy and safety of carrelizumab plus concurrent chemoradiotherapy compared with placebo plus concurrent chemoradiotherapy in the treatment of patients with inoperably advanced esophageal cancer, and to explore the relationship between PD-L1 expression and efficacy in tumor tissues. Experimental group: carrelizumab in combination with concurrent chemoradiotherapy PD-1: carrelizumab: 200 mg/3W Chemotherapy: Paclitaxel: 50 mg/m2/W Cisplatin: 25mg/m2/W Radiotherapy: 50.4 Gy / 28 f Chemotherapy drugs are used for 5 cycles, and carrelibizumab is used for up to 24 months until PD or is intolerable Control group: placebo-resistant in combination with chemoradiotherapy placebo: 200 mg/3 W Chemotherapy: Paclitaxel: 50 mg/m2/W Cisplatin: 25mg/m2/W Radiotherapy: 50.4 Gy / 28 f Chemotherapy drugs are used for 5 cycles, and carrelibizumab is used for up to 24 months until PD or is intolerable

DETAILED DESCRIPTION:
Experimental group: carrelizumab in combination with concurrent chemoradiotherapy PD-1: carrelizumab: 200 mg/3W Chemotherapy: Paclitaxel: 50 mg/m2/W Cisplatin: 25mg/m2/W Radiotherapy: 50.4 Gy / 28 f Chemotherapy drugs are used for 5 cycles, and carrelibizumab is used for up to 24 months until PD or is intolerable Control group: placebo-resistant in combination with chemoradiotherapy placebo: 200 mg/3 W Chemotherapy: Paclitaxel: 50 mg/m2/W Cisplatin: 25mg/m2/W Radiotherapy: 50.4 Gy / 28 f Chemotherapy drugs are used for 5 cycles, and carrelibizumab is used for up to 24 months until PD or is intolerable

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study and sign informed consent;
2. Age 18-75 years, including 18 and 75 years old, male or female;
3. Patients with histologically confirmed locally advanced esophageal squamous cell carcinoma with a clinical stage of stage II-IVa that is inoperably resectable (including unresectable, or has contraindications to surgery or refuses surgery) (according to the 8th edition AJCC stage, the pre-treatment clinical stage is: cT1N2-3M0, cT2-4bN0-3M0);
4. the presence of measurable and/or non-measurable lesions that meet the definition of the Efficacy Evaluation Criteria for Solid Tumors (RECIST1.1);
5. Have not received systemic antineoplastic therapy (including but not limited to systemic chemotherapy, molecularly targeted therapy, immunotherapy, biological therapy, topical therapy, and other investigational therapies)
6. ECOG: 0~1 point
7. Fresh or archived tumor tissue samples within 6 months (fresh samples preferred) must be provided for biomarker (such as PD-L1) analysis, the sample type is FFPE tumor tissue block or at least 5 unstained, 3-5 μm thick FFPE tumor tissue section, for subjects who cannot provide tissue samples that meet the above requirements, they can discuss with the sponsor to determine whether to enroll;
8. Expected survival≥ 3 months;
9. The function of vital organs meets the following requirements (no blood components and cell growth factors are allowed 2 weeks before starting screening tests):

   1. Absolute neutrophil count (ANC) ≥1.5×109/L;
   2. platelets≥ 100×109/L;
   3. hemoglobin≥ 9g/dL;
   4. serum albumin≥ 2.8 g/dL;
   5. Total bilirubin ≤ 1.5 × ULN, ALT, AST and/or AKP≤2.5 × ULN;
   6. Serum creatinine ≤1.5 × ULN or creatinine clearance ≥ 60 mL/min (calculated according to the Cockcroft-Gault formula, see Annex II);
   7. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5× ULN (can be screened for anticoagulation at a stable dose such as low molecular weight heparin or warfarin and INR within the expected therapeutic range of anticoagulants);
10. Female subjects of childbearing potential should have a urine or serum pregnancy test within 72 hours prior to receiving the first study drug administration and demonstrate a negative testament,and be willing to use an effective method of contraception during the trial period to 3 months after the last dose. For male participants whose partner is a woman of childbearing age, effective methods of contraception should be used during the trial and up to three months after the last dose

Exclusion Criteria:

1. history of surgery for esophageal cancer;
2. history of previous fistula due to primary tumor invasion;
3. a higher risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation;
4. participants with poor nutritional status with a BMI of less than 18.5 kg/m2 or a PG-SGA score of ≥9;
5. have undergone major surgery or severe trauma within 4 weeks prior to the first use of the study drug;
6. presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
7. Have received or are currently receiving any of the following treatments:

   1. Anti-PD-1 or anti-PD-L1 antibody therapy, chemotherapy, radiotherapy, targeted therapy;
   2. Have received any investigational drug within 4 weeks prior to the first use of the investigational drug;
   3. Participants who require systemic therapy with corticosteroids (> 10 mg prednisone equivalent per day) or other immunosuppressants within 2 weeks prior to the first study drug, except for local inflammation of the esophagus and for the prevention of allergies and nausea and vomiting. In other special circumstances, it is necessary to communicate with the sponsor. In the absence of active autoimmune disease, inhaled or topical steroid replacement and adrenocorticosteroid replacement at a dose > a potent dose of 10 mg/day prednisone is allowed;
   4. Those who have received an antitumor vaccine or have received a live vaccine within 4 weeks prior to the first dose of the study drug
8. have any active autoimmune disease or history of autoimmune disease (eg, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary physitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism); Except vitiligo or patients with asthma/allergies of the same age who have recovered and do not require any intervention in adulthood; Patients with autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone and type I diabetes mellitus treated with stable doses of insulin may be included;
9. a history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency disorders, or a history of organ transplantation and allogeneic bone marrow transplantation;
10. Subjects with uncontrolled cardiac clinical symptoms or diseases, such as (1) heart failure with NYHA II and above, (2) unstable angina, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
11. Severe infection (CTC AE> grade 2) within 4 weeks prior to the first use of the study drug, such as severe pneumonia, bacteremia, infection comorbidities, etc. requiring hospitalization; Baseline chest imaging suggests active lung inflammation, signs and symptoms of infection present in the 2 weeks prior to first study drug use requiring oral or intravenous antibiotic therapy, except for prophylactic antibiotics;
12. history of interstitial lung disease, noninfectious pneumonia, pulmonary fibrosis, or other uncontrolled acute lung disease;
13. Patients with active tuberculosis infection detected by history or CT examination, or patients with a history of active tuberculosis infection within 1 year prior to enrollment, or patients with a history of active tuberculosis infection more than 1 year before that have not been formally treated;
14. Participants had active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibodies and HCV-RNA above the lower limit of the assay);
15. Laboratory values of sodium, potassium, and calcium greater than grade 1 were abnormal in the first 2 weeks of randomization and could not be improved after treatment;
16. known allergy to macromolecular protein preparations, or to any carrelizul component, or allergy, hypersensitivity or contraindication to paclitaxel or cisplatin or any of the ingredients used in their preparations;
17. Any other malignancy diagnosed prior to the first use of the study drug, except for malignancies with a low risk of metastasis and death (5-year survival >90%), such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ;
18. pregnant or lactating women; participants of childbearing potential who are unwilling or unable to use effective contraception;
19. According to the investigator's judgment, the subject has other factors that may cause him to be forced to terminate the study halfway, such as other serious diseases (including psychiatric diseases) that require combined treatment, recent combination with other serious diseases (such as myocardial infarction, cerebrovascular accident) considering a high risk of recurrence, serious abnormal laboratory test values, family or social factors, which may affect the safety of subjects or the collection of trial data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
PFS evaluated by IRC | up to 2 years
  IRC stands for Independent Review Committee Assessment，Progression-free disease as assessed by an independent review committee Progression-free survival refers to the time from randomization to the first occurrence of disease progression or death from any cause

SECONDARY OUTCOMES:
OS Overall Survival | up to 2 years
  Overall survival was measured from the initiation of chemotherapy to the date of the last follow-up or death.
ORR | through study completion, an average of 18 month
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission
Progression-free survival evaluated by Researchers | up to 2 years
  The PFS was calculated from the initiation of chemotherapy to the date of disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin MM GE, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No